CLINICAL TRIAL: NCT05368740
Title: Evaluation of Thoracic Surgery Patients With Integrated Pulmonary Index: A Prospective, Observational Study
Brief Title: Integrated Pulmonary Index Monitoring for Thoracic Surgery Patients
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, associate professor, Cukurova University
Other Study IDs: IPI
Record Dates: First submitted 2022-04-22; First posted 2022-05-10 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Complications; Monitoring
Keywords: monitoring; postoperative complications; thoracic surgery; integrated pulmonary index
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- median IPI group: IPI score level was between 5-7
  Interventions: Device: integrated pulmonary index monitor
- high IPI group: IPI score level was between 8-10
  Interventions: Device: integrated pulmonary index monitor

INTERVENTIONS:
Device: integrated pulmonary index monitor — Integrated Pulmonary Index (IPI) is a new monitoring method calculated using respiratory rate (RR), end-tidal carbon dioxide (EtCO2), peripheral oxygen saturation (SpO2), and heart rate (HR). It is designed to obtain information about the patients' oxygenation and ventilation in the form of a single value or waveform from 1 to 10 with a mathematical algorithm using fuzzy logic. According to this scoring system; 10= normal, 8-9= within normal range, 7= close to normal range, requires attention, 5-6= requires attention and may require intervention, 3-4= requires intervention, 1-2= requires immediate intervention [2].
  Other Names: Capnostream-20, Medtronic

SUMMARY:
The aim of this study was to investigate the effect of postoperative Integrated Pulmonary Index (IPI) scores on postoperative complications, blood gas analysis, mortality and morbidity in the patients undergoing thoracic surgery.

DETAILED DESCRIPTION:
This prospective observational clinical study was performed between August 1, 2020 and January 31, 2021. After faculty ethics committee approval (Cukurova University, decision number: 111, date 02.10.2020) and written informed patient consent, 97 patients with American Society of Anesthesiologists (ASA) physical status I-II, over 18 years, volunteer to participate study, scheduled for elective VATS and thoracotomy surgery under general anesthesia were included in this study. Exclusion criteria were the presence of neuromuscular disorder, serious respiratory, cardiovascular, renal, and hepatic disease, ASA score > II, pneumonectomy surgery, morbid obesity with body mass index (BMI) > 40 kg/m2, younger than 18 years old, pre-determined need for postoperative intensive care.

Routine monitoring (electrocardiogram, noninvasive arterial blood pressure, heart rate and oxygen saturation) were applied before the induction of anesthesia to all patients. The induction was with intravenously (iv) 1.5-2 mg/kg propofol and 0.6 mg/kg rocuronium. After adequate muscle relaxation, female patients were intubated with a 35-37 F, male patients were intubated with a 39-41 F double-lumen tube. Anesthesia was maintained by repeated rocuronium doses if needed, 1.5-2% sevoflurane and an oxygen-air mixture. One lung ventilation was started just before the thorax was opened.

At the end of the surgery, neuromuscular block was antagonised with neostigmine (0.05 mg/kg) and atropine (0.015 mg/kg). Following extubation, patients were brought to the postanesthetic care unit (PACU) for 2 hours. For postoperative analgesia, regional techniques were used if the patients agreed, otherwise, iv opioid and nonsteroidal anti-inflammatory drugs (NSAIDs) were applied. All patients were given 2 L/minute oxygen as a standard with a nasal cannula. Postoperative pain was assessed by Visual Analog Scale (VAS), if the patients complained of pain (VAS ≥ 4), iv 0.5 mg/kg meperidine was given as a rescue analgesia.

Age, height, body weight, BMI, ASA physical status, comorbidity, and respiratory function test values were recorded as demographic data. Surgery type, duration of anesthesia, duration of surgery, and complications also were recorded. Systolic, diastolic, and mean blood pressure, SpO2, EtCO2, IPI values (monitored with the CapnostreamTM35 portable respiratory monitor), and arterial blood gas analyzes (evaluated with the ABL800 BASIC blood gas device) were recorded at the 15, 30, 60 and 120th minutes at the PACU. After 2 hours, when patients met standard PACU discharge criteria (fully awake, stable hemodynamic and respiratory parameters, satisfaction analgesia) they were transferred to the thoracic surgery ward.

All patients were evaluated in three groups according to their IPI score: high IPI (score level 8-10) group, medium IPI (score level 5-7) group, and low IPI (score level 1-4) group. Required attention was defined as SpO2 was between 88% and 92%, RR ≤ 8 breath/minute or IPI score level was between 5 and 7. The required intervention was defined as SpO2 ≤ 88% and IPI score level was ≤ 4. Postoperatively, at 6, 12, 18 and 24th hours, hemodynamic values and arterial blood gas analyses, length of hospital stay, complications, need for intensive care and 28-day mortality were evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I-II,
2. Over 18 years,
3. Scheduled for elective VATS and thoracotomy surgery under general anesthesia

Exclusion Criteria:

1. Neuromuscular disorder,
2. Serious respiratory disease,
3. Serious cardiovascular disease,
4. Renal failure,
5. Hepatic failure,
6. ASA score > II,
7. Pneumonectomy surgery,
8. Morbid obesity with body mass index (BMI) > 40 kg/m2,
9. Younger than 18 years old,
10. Pre-determined need for postoperative intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years) with ASA physical status I-II class, volunteer to participate study, scheduled for elective thoracotomy and video-assisted thoracoscopic surgery (VATS) between August 1, 2020 and January 31, 2021 were included in our analysis.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
number of participants with postoperative complications | postoperative first 24 hours
  The patients were visited in the thoracic surgery service and postoperative complications were recorded.
arterial blood pH values in the first 24 hours postoperatively | postoperative first 24 hours
  The patients were visited in the thoracic surgery service, blood gas analyses were analysis and arterial blood pH values were recorded.

SECONDARY OUTCOMES:
length of hospital stay | through study completion, an average of 1 week"
  Postoperatively, the patients were visited in the thoracic surgery service everyday and length of hospital stay was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Mediha Türktan, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No